CLINICAL TRIAL: NCT04854252
Title: A Comparison of Opioid-containing Anesthesia Versus Opioid-free Anesthesia Using the Cortínez-Sepúlveda Model on Differential Cytokine Responses in Patients Undergoing Gastric Bypass Surgery
Brief Title: Inflammatory Response to Opioid Versus Opioid Free Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, ERIKA MARTINEZ-LOPEZ, PhD, University of Guadalajara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 09042021
Record Dates: First submitted 2021-04-11; First posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Morbid Obesity; Opioid Use; Fentanyl Adverse Reaction; Cytokine Storm
Keywords: Morbid obesity; Gastric bypass; Opioid containing anesthesia; Opioid free anesthesia; Cytokines
MeSH Terms: conditions — Obesity, Morbid; Cytokine Release Syndrome | interventions — Fentanyl

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to two anesthesia groups: opioid-containing (n=20) or opioid-free (n=20). The opioid used in the opioid-containing anesthesia group was fentanyl.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Inflammatory response to opioid vs opioid free anesthesia (Experimental): Patients were randomly assigned to two anesthesia groups: opioid-containing (n=20) or opioid-free (n=20). The opioid used in the opioid-containing anesthesia group was fentanyl.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — TIVA opioid-containing anesthesia: fentanyl in a bolus dose of l3 mcg/kg (corrected weight) TIVA opioid-free anesthesia: dexmedetomidine 1-1.5 mcg/kg (corrected weight) for 40 minutes

SUMMARY:
Anesthetic agents, including opioids can modulate the altered immune function in patients with obesity through mechanisms that involve the expression and release of cytokines. For this reason, anesthetic care in patients with obesity remains controversial. Therefore, the aim of the study was to compare the effect of opioid-containing anesthesia vs opioid-free anesthesia using the Cortínez-Sepúlveda model on serum levels of IL-6, IL-1β and TNF-α before and after surgery in obese patients undergoing bypass surgery.

Methods: A randomized cross-sectional study of 40 unrelated obese adults was performed in the Anesthesiology and Bariatric Surgery Service at the Civil Hospital of Guadalajara "Dr. Juan I. Menchaca". Before undergoing laparoscopic Roux-en-Y gastric bypass, patients were randomly assigned to two anesthesia groups: opiod-containing (n=20) or opioid-free (n=20). The opioid used in the opioid-containing anesthesia group was fentanyl. To characterize the disposition of intravenous propofol for the target-controlled infusion technique in obese patients, the Cortínez-Sepúlveda pharmacokinetic model was used. Body mass was determined to the nearest 0.05kg using a balance scale (Seca 703; Seca, Hamburg, Germany). Blood samples were taken before and immediately after surgery and cytokine serum levels were determined with ELISA kits. Statistical analyses were performed using the IBM Statistical Package for the Social Sciences software package version 20.0 (IBM Corp., Armonk, NY, USA).

ELIGIBILITY:
Inclusion Criteria:

* Who were scheduled for bypass surgery at the Service of Anesthesiology and Bariatric Surgery of the Civil Hospital of Guadalajara "Dr. Juan I Menchaca", Jalisco, Mexico, were recruited.

Exclusion Criteria:

* Patients with a history of ischemic heart disease, history of drug abuse, and with any known allergy to any of the drugs used during anesthesia. Elimination criteria were: patients who withdrew their consent or with insufficient and poor quality blood samples (coagulated) or other reasons that did not allow sample processing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

PRIMARY OUTCOMES:
Differences in the inflammatory response determined by serum cytokine levels when using opioid-containing anesthesia or opioid-free anesthesia in patients undergoing bypass surgery | 30 minutes before the anesthesia administration and 5 minutes before extubation
  Cytokine serum levels were measured with an enzyme-linked immunosorbent (ELISA) assay. LEGEND MAX™ Human IL-1β (cat # 437007), LEGEND MAX™ Human IL-6 (cat # 430507) and LEGEND MAX™ Human TNF-α (cat # 430207) ELISA kits

CONTACTS AND LOCATIONS:
Locations (1):
- Erika Martínez-López, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Campos-Perez W, Ramirez-Plascencia L, Perez-Robles M, Rivera-Valdes JJ, Sanchez-Munoz P, Perez-Vargas L, Gonzalez-Landeros D, Cuevas JHM, Martinez-Lopez E. A comparison of opioid-containing anesthesia versus opioid-free anesthesia using the Cortinez-Sepulveda model on differential cytokine responses in obese patients undergoing gastric bypass surgery: a randomized controlled trial. BMC Anesthesiol. 2022 Sep 16;22(1):294. doi: 10.1186/s12871-022-01838-8. PMID 36114460